CLINICAL TRIAL: NCT05017649
Title: Characterization of Adenosine A2A Receptor Expression and Fubnction in Hypercholesterolemic Patients
Brief Title: Role of A2A Receptor in Hypercholesterolemic Patients
Acronym: RASCAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-07; ID-RCB (Other: 2021-A01196-35)
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; adenosine receptor; PBMC
MeSH Terms: conditions — Hypercholesterolemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Other): volunteers showing no hypercholesterolemia
  Interventions: Biological: Blood sample
- Patients with untreated hypercholesterolemia at the time of inclusion (Experimental): patients presenting hypercholesterolemia with no treatment at the time of inclusion
  Interventions: Biological: Blood sample
- Patients with treated hypercholesterolemia at the time of inclusion (Experimental): patients presenting hypercholesterolemia and treated at the time of inclusion
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sampling.

SUMMARY:
Hypercholesterolemia promotes chronic inflammation, endothelial dysfunction, atherosclerosis and is a major risk factor for cardiovascular disease (CVD). Treatment with lipid-lowering drugs (statins, ezetimibe, PCSK9 inhibitors or LDL-apheresis) reduces the risk of major cardiovascular events in proportion to the absolute reduction of LDL-cholesterol (LDL-C). Nevertheless, a better understanding of the effects of hypercholesterolemia on the cardiovascular and immune systems could help identify all the mechanisms responsible for the excess risk of CVD in hypercholesterolemic patients and develop better prevention and treatment strategies.

Adenosine via A2A receptors (A2AR) plays a crucial role in the regulation of the cardiovascular and immune systems.

In this project, the investigators wish :

* To study whether the expression and function of A2AR in PBMCs are altered in human hypercholesterolemia, using as a study model a larger cohort of patients with hypercholesterolemia of increasing level and severity: polygenic form, heterozygous genetic form and homozygous genetic form in comparison with healthy subjects with normal cholesterol levels.
* To study whether A2AR expression and function in PBMCs are associated with blood levels of LDL-C and homocysteine and with the inflammatory status of patients.
* To assess whether the cholesterol-lowering therapies currently used to reduce LDL-C levels and thus the risk of CVD in hypercholesterolemic patients have an impact on possible alterations of A2AR expression and function in PBMCs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-80 years
* For the group of hypercholesterolemic patients :

  * LDL-cholesterol level >1.9 g/L with or without treatment to make the diagnosis of hypercholesterolemia (laboratory test less than 12 months old at inclusion)
* For the healthy group :

  ● No cholesterol-modifying therapy.
* Subject not having hypercholesterolemia (biological assessment less than 12 months old at inclusion with LDL-cholesterol level < 1.9 g/L) and not taking cholesterol-lowering treatment.
* Subjects who are affiliated or beneficiaries of a social security plan
* Subject agreeing to participate in the study and having signed an informed consent

Exclusion Criteria:

* Protected person, as defined by articles L1121-5, L1121-6 and L1121-8 of the Public Health Code: pregnant or breastfeeding woman, person deprived of liberty by judicial decision, adult person unable to give consent.
* Person who does not understand the French language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Quantification of A2AR expression in PBMCs | Baseline
  Comparison between hypercholesterolemic patients and healthy volunteers
Quantification of A2AR expression in PBMCs | 3 months after initiation of treatment
  Comparison between hypercholesterolemic patients and healthy volunteers
Quantification of A2AR function in PBMC | 3 months after initiation of treatment
  Comparison between hypercholesterolemic patients and healthy volunteers
Quantification of A2AR function in PBMC | Baseline
  Comparison between hypercholesterolemic patients and healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — AP-HM
Locations (1):
- Service Endocrinologie, Marseille, France

IPD SHARING:
Plan to Share IPD: No